CLINICAL TRIAL: NCT03889756
Title: Ketamine for Severe Adolescent Depression: Intermediate-term Safety and Efficacy
Acronym: SAD-KIDS
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: No more funding available to continue since we could not recruit throughout the pandemic.
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2000023857
Record Dates: First submitted 2019-03-22; First posted 2019-03-26 (Actual); Results first posted 2023-04-24 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2023-03

CONDITIONS: Major Depressive Disorder
Keywords: depression, ketamine
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Intervention Model Description: Phase 1 is a double-blind, midazolam-controlled parallel design trial; Phase 2 is an open extension.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will not be told what medication they are receiving; physicians absent from the infusion paradigm will perform blinded clinical efficacy ratings.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ketamine (Experimental): Ketamine is an FDA-approved anesthetic agent that is commonly used to induce surgical anesthesia due to its low incidence of significant respiratory depression and hypotension. It as a N-methyl-D-aspartate (NMDA) receptor antagonist and glutamatergic modulator, and has been demonstrated in multiple controlled clinical trials to have rapidly acting antidepressant and anti-suicidal effects in adults.
  Interventions: Drug: Ketamine infusion
- Midazolam (Placebo Comparator): Midazolam, the active control in this study, is a medication that is approved by the Food and Drug Administration as a sedative for both children and adults.It is a benzodiazepine with a short half-life that was chosen so as to blind the psychotomimetic effects of Ketamine.
  Interventions: Drug: Midazolam infusion

INTERVENTIONS:
Drug: Ketamine infusion — The dose of ketamine established in prior research (0.5 mg/kg over 40 minutes) will be used in this study to minimize risks. The maximum total single dose allowed in this study will be 40mg, corresponding to a weight of 80kg.
  Arms: Ketamine
Drug: Midazolam infusion — The weight-based midazolam dosing established in prior ketamine trials in adults (0.045mg/kg) will be used to minimize risks, as this is considered a very low dose compared to the sedation literature. The maximum total dose allowed in this study will be 3.6mg per infusion, corresponding to a weight of 80kg.
  Arms: Midazolam

SUMMARY:
The purpose of this study is to evaluate the intermediate-term efficacy and tolerability of a multiple-dosing ketamine infusion paradigm for the treatment of medication-refractory major depressive disorder (MDD). We are using a two-phase design. The first phase is a 3-week double blind parallel design clinical trial comparing 6 infusions of ketamine compared to 6 infusions of midazolam in 24 adolescents with treatment resistant depression. The primary outcome of this phase will be Children's Depression Rating Scale (CDRS) score at Day 18. The second phase is a 6-month open phase in which patients who received midazolam and remain depressed with be offered open ketamine treatment (6 infusions over 3 weeks). All participants will be followed weekly for 6 months and tracked for time to relapse.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the intermediate-term efficacy and tolerability of a multiple-dosing ketamine infusion paradigm for the treatment of medication-refractory major depressive disorder (MDD). The specific aims of the study are: To evaluate the efficacy and tolerability of a multiple-dosing ketamine infusion paradigm (2 infusions per week for 3 weeks) compared to midazolam in adolescents with treatment resistant depression (TRD), . To test these aims we have designed a two-phase trial. The first phase is a 3-week double blind parallel design clinical trial comparing 6 infusions of ketamine compared to 6 infusions of midazolam in 24 adolescents with TRD. The primary outcome of this phase will be Children's Depression Rating Scale (CDRS) score at Day 18. The second phase is a 6-month open phase in which patients who received midazolam and remain depressed with be offered open ketamine treatment (6 infusions over 3 weeks). All participants will be followed weekly for 6 months and tracked for time to relapse. In those who initially responded to ketamine, symptom triggered maintenance infusions will be offered during this 6-month time period. All participants will receive standard of care treatment in addition to experimental procedures, and will be tracked monthly with extensive neurocognitive assessments.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ages 13-17 years
2. Meet DSM-5 (Diagnostic and Statistical Manual 5 ) criteria for Major Depressive Disorder by structured interview (MINI-KID)
3. Children's Depression Rating Scale, Revised CDRS score ≥40 at screening
4. Failure to achieve remission with at least 2 antidepressant trials (e.g. SSRI, SNRI or TCA), meaning at least 6 weeks at therapeutic dosing, including at least 4 weeks of stable dosing
5. Stable psychiatric medications and doses for the month prior to enrollment. Subjects may continue to engage in any ongoing psychotherapy.
6. Medically and neurologically healthy on the basis of physical examination and medical history.
7. Parents able to provide written informed consent and adolescents must additionally provide assent.

Exclusion Criteria:

1. History of psychotic disorder, manic episode, autism spectrum disorder diagnosed by MINI-KID
2. History of substance dependence diagnosis by MINI-KID (excluding tobacco) or positive urine toxicology.
3. Intellectual disability (IQ<70) per medical history
4. Pregnancy (urine pregnancy tests on the day of infusions for menstruating girls) or lactation
5. Prior treatment with ketamine for depression or prior recreational use of ketamine.
6. Inability to provide written informed consent according to the Yale Human Investigation Committee (HIC) guidelines in English.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3 (Actual)
Dates: Start 2019-07-17 (Actual); Primary Completion 2019-12-18 (Actual); Study Completion 2023-01-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael H. Bloch, MD, Principal Investigator — Yale University; Jennifer Dwyer, MD, Study Director — Yale University
Locations (1):
- Yale Child Study Center, New Haven, Connecticut, United States

REFERENCES:
- [Background] Richmond TK, Rosen DS. The treatment of adolescent depression in the era of the black box warning. Curr Opin Pediatr. 2005 Aug;17(4):466-72. doi: 10.1097/01.mop.0000166347.53102.e7. PMID 16012257
- [Background] Krystal JH, Karper LP, Seibyl JP, Freeman GK, Delaney R, Bremner JD, Heninger GR, Bowers MB Jr, Charney DS. Subanesthetic effects of the noncompetitive NMDA antagonist, ketamine, in humans. Psychotomimetic, perceptual, cognitive, and neuroendocrine responses. Arch Gen Psychiatry. 1994 Mar;51(3):199-214. doi: 10.1001/archpsyc.1994.03950030035004. PMID 8122957
- [Background] Zarate CA Jr, Singh JB, Carlson PJ, Brutsche NE, Ameli R, Luckenbaugh DA, Charney DS, Manji HK. A randomized trial of an N-methyl-D-aspartate antagonist in treatment-resistant major depression. Arch Gen Psychiatry. 2006 Aug;63(8):856-64. doi: 10.1001/archpsyc.63.8.856. PMID 16894061
- [Background] Murrough JW, Iosifescu DV, Chang LC, Al Jurdi RK, Green CE, Perez AM, Iqbal S, Pillemer S, Foulkes A, Shah A, Charney DS, Mathew SJ. Antidepressant efficacy of ketamine in treatment-resistant major depression: a two-site randomized controlled trial. Am J Psychiatry. 2013 Oct;170(10):1134-42. doi: 10.1176/appi.ajp.2013.13030392. PMID 23982301
- [Background] Wilkinson ST, Toprak M, Turner MS, Levine SP, Katz RB, Sanacora G. A Survey of the Clinical, Off-Label Use of Ketamine as a Treatment for Psychiatric Disorders. Am J Psychiatry. 2017 Jul 1;174(7):695-696. doi: 10.1176/appi.ajp.2017.17020239. No abstract available. PMID 28669202

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ketamine | Midazolam
Started | 1 | 2
Completed | 1 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Demographic data will be presented together to avoid unblinding of subjects due to small number of participants
Groups:
- Overall Participants: Participants enrolled in the trial. Due to the small sample size, data will be presented together to avoid unblinding.
Arm/Group | Overall Participants
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] — Age at the time of enrollment to the trial.
  years | 16.3 [16 to 17]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of a Multiple-dosing Ketamine Infusion Paradigm (2 Infusions Per Week for 3 Weeks) Compared to Midazolam in Adolescents With Treatment Resistant Depression Using the Children's Depression Rating Scale (CDRS)
Description: Establish if repeated ketamine will be efficacious medically and psychiatrically, as measured by a significant reduction in CDRS score in those treated with ketamine at the end of the dosing paradigm. The Children's Depression Rating Scale (CDRS) is a clinician-rated instrument with 17 items scored on a 1 to 5 or 1 to 7 scale. A rating of 1 indicates normal, thus the minimum score is 17. The maximum score is 113. Scores of 20-30 suggest borderline depression. Scores of 40-60 indicate moderate depression.
Time Frame: Day 18
Population: all those enrolled in the study prior to termination
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Ketamine | Midazolam
Number analyzed (Participants) | 1 | 2
score on a scale | 42 [42 to 42] | 62 [62 to 62]

2. Primary Outcome: Tolerability of a Multiple-dosing Ketamine Infusion Paradigm (2 Infusions Per Week for 3 Weeks) Compared to Midazolam in Adolescents With Treatment Resistant Depression
Description: Establish if repeated ketamine will be tolerated as measured by drop-out counts.
Time Frame: Day 18
Measure: Count of Participants; unit: Participants
Arm/Group | Ketamine | Midazolam
Number analyzed (Participants) | 1 | 2
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 6 months
Arm/Group | Ketamine | Midazolam
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/2
Other Adverse Events (participants affected / at risk) | 1/1 | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ketamine (N=1) | Midazolam (N=2)
Diplopia (Eye disorders) | 1 | 2
Numbness (Nervous system disorders) | 1 | 2
Blurred Vision (Eye disorders) | 1 | 2
Dizziness (Nervous system disorders) | 1 | 2
Tachycardia (Cardiac disorders) | 1 | 1
Headache (Nervous system disorders) | 1 | 2
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 2
Palpitations (Cardiac disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hearing Changes (Ear and labyrinth disorders) | 1 | 0
Pruritus at Infusion Site (Skin and subcutaneous tissue disorders) | 1 | 0
Tics (Nervous system disorders) | 1 | 0
Lightheadedness (Nervous system disorders) | 1 | 0
Joint Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Stress Fracture (Musculoskeletal and connective tissue disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
The study was only able to enroll 3 participants before the pandemic started and then ran out of funding to finish the trial. Presented are summary data and to avoid revealing any identifying information of participants, data is presented overall where applicable (e.g. baseline characteristics).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-03): https://cdn.clinicaltrials.gov/large-docs/56/NCT03889756/Prot_SAP_000.pdf